CLINICAL TRIAL: NCT05609006
Title: Compliance With a High Energy Content, Low Volume Oral Nutritional Supplement (ONS)
Brief Title: Compliance With a High Energy Content, Low Volume Oral Nutritional Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Specialized Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NUT 2.4 Study
Record Dates: First submitted 2022-10-31; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: High-Energy, Low-Volume ONS // High-Energy Standard ONS (Experimental): Intervention: high-energy low-volume ONS (2.4kcal/ml; 125ml) for 28 days followed by high-energy standard ONS (2.0kcal/ml; 200ml) for 28 days
  Interventions: Dietary Supplement: High-Energy, Low-Volume ONS; Dietary Supplement: High-Energy Standard ONS
- Group B: High-Energy Standard ONS // High-Energy, Low-Volume ONS (Experimental): Intervention: high-energy standard ONS (2.0kcal/ml; 200ml) for 28 days followed by high-energy low-volume ONS (2.4kcal/ml; 125ml) for 28 days
  Interventions: Dietary Supplement: High-Energy, Low-Volume ONS; Dietary Supplement: High-Energy Standard ONS

INTERVENTIONS:
Dietary Supplement: High-Energy, Low-Volume ONS — 2 bottles/day of a High-Energy, Low-Volume ONS
  Other Names: Energy-dense ONS; 2.4 ONS
Dietary Supplement: High-Energy Standard ONS — 2 bottles/day of a High-Energy Standard ONS
  Other Names: 2.0 ONS

SUMMARY:
This study aims to investigate the compliance of high-energy, low-volume oral nutritional supplements (ONS) compared to equivalent high-energy standard ONS (control) in participants at risk of malnutrition.

DETAILED DESCRIPTION:
The use of high-calorie, high-protein ONS is recommended in patients with malnutrition or who are at risk of malnutrition-related disease. However, compliance with ONS is a key feature to improve the patient's nutritional status. Since compliance with ONS could be influenced by the energy density and the volume of the nutritional supplement used, a higher energy density and lower volume ONS could provide similar energy to the standard ONS for the requirements of this population.

This study has been designed as an open-label randomized crossover study with nutritional intervention with the aim to compare the patient's compliance, defined as the percentage of energy consumed with respect to that prescribed, with a high-energy content, low volume ONS versus a standard high calorie and volume ONS, over an 8-weeks follow-up period. As secondary objectives, the study aims to describe the gastrointestinal tolerance and satisfaction of the study ONS, to establish the factors that may affect compliance with the ONS and to compare the cost associated with product wastage in both ONS.

The study population will consist of patients aged ≥ 18 years, distributed into three groups according to their diagnosis: oncological patients, surgical patients, and other patients, all of them malnourished or at risk of malnutrition according to Subjective Global Assessment (SGA), and requiring the use of an ONS. Participants will be randomly allocated to receive either:

Group A: A high energy, low volume ONS (2.4kcal/ml; 125ml) in addition to the diet for 28 days. Participants will then receive the equivalent standard ONS (2.0kcal/ml, 200ml) as control ad libitum in addition to diet for 7 days, or:

Group B. A standard ONS (2.0 kcal/ml, 200ml) as control in addition to the diet for 28 days. Participants will then receive the high energy, low volume equivalent ONS (2.4kcal/ml; 125ml) for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Patients who are in one of the following clinical situations: oncological patients who did not undergo surgery during the month prior to inclusion, including head and neck, esophagus, stomach, pancreas, or colon cancer; surgical patients who underwent surgery less than one month, including all types of surgical processes; and other non-surgical patients diagnosed with benign esophageal stricture, chronic radiation enteritis, and non-oncological maxillofacial pathology, cystic fibrosis, human immunodeficiency virus (HIV), malabsorption syndrome , ulcerative colitis, Crohn's disease, fistula, intestinal pseudo-obstruction, chronic obstructive pulmonary disease (COPD), congestive heart failure (CHF), or who were undergone to scheduled major surgery or transplantation within a period of no less than 2 months until inclusion.
* Patients with malnutrition or at risk of malnutrition according to Subjective Global Assessment (SGA).
* Patients with a high energy requirement that require 2 bottles/day of an ONS (≥2kcal/ml), for a minimum period of 8 weeks
* Patients who have not received ONS during the month prior to their inclusion. Surgical patients may have received ONS prior to the study in accordance with the guidelines of the institution.
* Patients who voluntarily agree to participate in the study and give their signed consent for participation.

Exclusion Criteria:

* Patients suffering from any of the following clinical disorders: chronic kidney insufficiency or diabetes.
* Patients requiring enteral tube feeding or parenteral nutrition.
* Patients suffering from an allergy or intolerance to the product ingredients.
* Patients scheduled for surgery during the study period.
* Patients who, in the opinion of the treating physician, are unable to adhere to the protocol instructions, including inability of the patient/caregiver to use the study eCRF, and to remain in the study during all the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Compliance rate with ONS | One period of 28 days for both ONS (high-energy low-volume, and high-energy standard)
  Percentage of consumed energy over the prescribed

SECONDARY OUTCOMES:
Gastrointestinal tolerance | Weekly (from second to fourth week of each period) up to 8 weeks
  Tolerance is measured using a numeric rate scale (NRS) of the frequency of symptoms (0, not at all; 10, very frequently) for the last 7 days such as nausea, vomiting, diarrhea, constipation, acid reflux, bellyache, bloated belly, stomach pain, flatulence, and satiety.
Satisfaction with ONS | For each period/ONS, up to 8 weeks
  Satisfaction with the ONS taste, satiety, ease of completing the intake, and overall satisfaction are measured using an NRS of the level of satisfaction (0, very dissatisfied; 10, very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Leon, MD, Principal Investigator — Hospital Universitario 12 de Octubre; Gabriel Olveira, MD, Principal Investigator — Hospital Regional de Malaga
Locations (2):
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Málaga, Málaga

IPD SHARING:
Plan to Share IPD: No